CLINICAL TRIAL: NCT07025031
Title: Maternal Serum Progesterone And Placental Heme Oxgenase-1 Expression In Early Onset Idiopathic Fetal Growth Restriction: A Case Control Study
Brief Title: Fetal Growth Restriction a Case Control Study
Status: Not yet recruiting | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Other Study IDs: JEP-2025-183
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Fetal Growth Restriction
Keywords: progesterone; Heme Oxygenase-1; Idiopathic fetal growth restriction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal blood Placenta
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with pregnancies affected by idiopathic fetal growth restriction: Women with normal pregnancies and normally growing foetus

SUMMARY:
The study aims to investigate the responsible factors that leads to idiopathic fetal growth restriction.

DETAILED DESCRIPTION:
The study aims to investigate the relationship between maternal serum level of progesterone, immune-expression of HMOX-1 a placental angiogenesis marker with idiopathic fetal growth restriction.

ELIGIBILITY:
Inclusion Criteria:

* singleton
* dated pregnancy

Exclusion Criteria:

* fetus with structural or chromosomal anomaly
* receive treatments such as aspirin, progestogen, low molecular weight heparin
* has pre-existing medical disorders such as autoimmune disease, hypertension, diabetes
* smoking
* suspected intrauterine infection

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Study Population: Women diagnosed to have fetal growth restriction within 24 until 32 weeks gestation the absence of hypertension, diabetes or autoimmune disease.
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Maternal serum level of progesterone | At the point of recruitment from 24 until 32 weeks gestation.
  Maternal blood will be withdrawn and serum isolated. Measurement of progesterone level will be performed from the serum sample using ELISA.
Placental immunoexpression of Heme Oxygenase 1 | At delivery within 24 until 38 weeks gestation.
  Immunoexpression of Heme Oxygenase 1 in syncytiotrophoblasts, cytotrophoblasts, fetal endothelial cells, maternal vessels and decidual cells.

SECONDARY OUTCOMES:
Placenta histopathology examination | At delivery within 24 until 38 weeks gestation
  Placenta will be examined histopathologically

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared if necessary